CLINICAL TRIAL: NCT03590379
Title: A Phase II, Multicentre, Randomised, Double-blind, Double-dummy, Active-controlled, 3-way Cross-over Study to Evaluate the Efficacy of CHF 5993 Administered Via Dry Powder Inhaler (DPI) Versus CHF 5993 Via Pressurized Metered Dose Inhaler (pMDI) and CHF 1535 pMDI in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of Fixed Combination of Beclomethasone Dipropionate (BDP) + Formoterol Fumarate (FF) + Glycopyrronium Bromide (GB) (CHF 5993)Administered Via Dry Powder Inhaler (DPI) in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: TRI-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-05993BA1-02; 2017-004405-41 (EudraCT Number)
Record Dates: First submitted 2018-06-06; First posted 2018-07-18 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHF 5993 DPI (Experimental): BDP/FF/GB DPI 100/6/12,5 mcg
  Interventions: Drug: CHF 5993 DPI; Drug: Placebo pMDI
- CHF 5993 pMDI (Active Comparator): BDP/FF/GB pMDI 100/6/12,5 mcg
  Interventions: Drug: CHF5993 pMDI; Drug: Placebo DPI
- CHF 1535 pMDI (Active Comparator): BDP/FF pMDI 100/6 mcg
  Interventions: Drug: CHF 1535 pMDI; Drug: Placebo DPI

INTERVENTIONS:
Drug: CHF 5993 DPI — BDP/FF/GB DPI
  Arms: CHF 5993 DPI
Drug: CHF5993 pMDI — BDP/FF/GB pMDI
  Arms: CHF 5993 pMDI
Drug: CHF 1535 pMDI — BDP/FF pMDI
  Arms: CHF 1535 pMDI
Drug: Placebo DPI — CHF 5993 DPI matched placebo
  Arms: CHF 1535 pMDI; CHF 5993 pMDI
Drug: Placebo pMDI — CHF 5993 pMDI matched Placebo (direct blinding of active CHF 5993 and CHF 1535 pMDIs)
  Arms: CHF 5993 DPI

SUMMARY:
The purpose of this study is to evaluate the efficacy of Fixed Combination of Beclomethasone Dipropionate + Formoterol Fumarate + Glycopyrronium Bromide Administered Via Dry Powder Inhaler in COPD

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (40 ≤ age ≤ 85 years) with a diagnosis of COPD;
* Current smokers or ex-smokers;
* A Post-bronchodilator FEV1 ≥30% and <80% of the predicted normal value and FEV1/FVC (Forced Vital Capacity) < 0.7;
* Patients' COPD therapy (stable regimen at least 30 days before screening) with either:

  * Inhaled corticosteroids/long-acting β2-agonist/long-acting muscarinic antagonist (free or fixed) combination
  * Inhaled corticosteroids/long-acting β2-agonist (free or fixed) combination
  * Inhaled long-acting β2-agonist/long-acting muscarinic antagonist (free or fixed) combination
  * Inhaled long-acting muscarinic antagonist alone.

Exclusion Criteria:

* Pregnant and lactating women;
* Diagnosis of asthma;
* Known respiratory disorders other than COPD;
* Patients treated for a moderate or severe COPD exacerbation within 6 weeks prior to screening or during the run-in period;
* Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia;
* Patients who have clinically significant cardiovascular condition;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-12h (Area Under the Curve for Forced Expiratory Volume in 1 second measured serially for 0-12 hours) normalised by time (L) on dosing Day 28 | Day 28
  To demonstrate the non-inferiority between CHF 5993 DPI and CHF 5993 pMDI in terms of FEV1 AUC0-12h normalized by time, in COPD patients
Trough FEV1 at 24 hours (L) on dosing Day 28. | Day 28
  To demonstrate the non-inferiority between CHF 5993 DPI and CHF 5993 pMDI in terms of trough FEV1 at 24h on dosing Day 28 in COPD patients

SECONDARY OUTCOMES:
Change from baseline in pre-dose morning FEV1 (L) on Day 28 | from Baseline to Day 28
  To evaluate the efficacy of CHF 5993 DPI on other lung function parameters and clinical outcome measures.
Change from baseline in FEV1 AUC0-4h normalised by time (L) on Day 28 | from Baseline to Day 28
  To evaluate the efficacy of CHF 5993 DPI on other lung function parameters and clinical outcome measures.
Change from baseline in FEV1 AUC0-12h normalised by time (L) on Day 1 | from Baseline to Day 1
  To evaluate the efficacy of CHF 5993 DPI on other lung function parameters and clinical outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Michael Beeh, MD, Principal Investigator — Institut fuer Atemwegsforschung GmbH, Wiesbaden, Germany
Locations (1):
- Medical Center Convex EOOD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Result] Beeh KM, Kuna P, Corradi M, Viaud I, Guasconi A, Georges G. Comparison of Dry-Powder Inhaler and Pressurized Metered-Dose Inhaler Formulations of Extrafine Beclomethasone Dipropionate/Formoterol Fumarate/Glycopyrronium in Patients with COPD: The TRI-D Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2021 Jan 14;16:79-89. doi: 10.2147/COPD.S291030. eCollection 2021. PMID 33488071
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2017-004405-41/results